CLINICAL TRIAL: NCT07187960
Title: Randomized, Open Label, Multicenter Phase III Clinical Trial Evaluating the Efficacy and Safety of TQB2825 Injection Compared to Immunotherapy in the Treatment of Relapsed/Refractory Follicular Lymphoma
Brief Title: Evaluation of the Efficacy and Safety of TQB2825 Injection Compared to Immunotherapy in the Treatment of Recurrent/Refractory Follicular Lymphoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Chia Tai Tianqing Pharmaceutical Technology Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQB2825-III-01
Record Dates: First submitted 2025-09-17; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-03

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Rituximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB2825 Injection (Experimental): TQB2825 single drug intravenous injection, 28 days as a treatment cycle.
  Interventions: Drug: TQB2825 Injection
- Rituximab Injection (Active Comparator): Rituximab combined with Chemotherapy regimen, 21 days as a treatment cycle.
  Interventions: Drug: Rituximab Injection

INTERVENTIONS:
Drug: TQB2825 Injection — TQB2825 is a Cluster of Differentiation 3 (CD3) × Cluster of Differentiation 20 (CD20) bispecific antibody.
  Arms: TQB2825 Injection
Drug: Rituximab Injection — Rituximab combined with Chemotherapy (Rituximab, Cyclophosphamide, doxorubicin, Vincristine, Prednisone, Ifosfamide, Gemcitabine, cisplatin, Carboplatin, Etoposide, MESNA, Dexamethasone)
  Arms: Rituximab Injection

SUMMARY:
Evaluation of the efficacy and safety of TQB2825 injection compared to immunotherapy in the treatment of recurrent/refractory follicular lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily join this study, sign the informed consent form (ICF), and have good compliance.
2. 18 years old ≤ age<80 years old (calculated based on the date of signing the informed consent form); No gender restrictions; Eastern Cooperative Oncology Group Performance Status (ECOG) score 0-2.
3. Expected survival is greater than 6 months.
4. Follicular lymphoma (histological grade 1-3a) that meets the 2016 WHO diagnostic criteria or classic follicular lymphoma that meets the 2022 World Health Organization (WHO) diagnostic criteria, and immunophenotyping analysis shows CD20 positivity in the tumor.
5. Relapsed/refractory diseases that have received at least 2 lines of systemic treatment (at least 1 line containing CD20 monoclonal antibody) in the past, and have progressed during the most recent treatment period or relapsed after completing treatment, or have been confirmed to have no objective remission after sufficient treatment.
6. According to the 2014 Lugano criteria, there is at least one measurable lesion, which is a lymph node lesion with a length diameter greater than 15 mm or an extranodal lesion with a length diameter greater than 10 mm based on CT cross-sectional imaging.
7. The organ function is good.
8. Women of childbearing age should agree to use effective contraception during the study period and for 12 months after the end of study treatment, and agree not to donate eggs (oocytes) for reproductive purposes during this period; Not allowed to be in lactation period and have a negative serum or urine pregnancy test within 7 days before enrollment; Male patients who have not undergone vasectomy and their fertile female partners should agree to use effective contraceptive measures during the study period until 12 months after the end of the study treatment, and agree not to donate sperm during this period.

Exclusion Criteria:

1. Have had or currently have other malignant tumors within the previous 5 years of randomization. The following two situations can be included in the group: other malignant tumors that have been cured by a single surgery and have achieved continuous disease-free survival (DFS) for 5 years; Cured cervical carcinoma in situ, non melanoma skin cancer, and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ), and T1 (tumor infiltrating basement membrane)].
2. Lymphoma has previously or currently affected or is suspected to affect the central nervous system, or there is evidence of lymphoma leukemia present.
3. There is evidence of transformation into diffuse large B-cell lymphoma or other types of lymphoma (such as biopsy showing large cells or Positron Emission Tomography (PET) showing significant abnormal high metabolism in one/some lymph nodes).
4. Active hepatitis or decompensated cirrhosis (Child Pugh liver function rating B or C). (Note: active hepatitis B refers to positive HBsAg, and Hepatitis B Virus (HBV) DNA is positive or the test value exceeds the upper limit of normal value; Active hepatitis C refers to Hepatitis B Virus (HCV) antibody positivity, and HCV RNA positivity or detection value exceeding the upper limit of normal; The eligible subjects with positive hepatitis B HBsAg but HBV DNA not exceeding the upper limit of normal value, whether their HBV DNA is measurable or not, need to continue antiviral treatment (nucleoside analogues are recommended) and regularly monitor HBV DNA; For subjects with positive hepatitis B HBcAb but negative HBsAg, HBV DNA needs to be monitored regularly, and preventive antiviral treatment is recommended; For subjects who are positive for hepatitis C HCV antibodies but whose HCV RNA does not exceed the upper limit of normal values, regular monitoring of HCV RNA is required.
5. The adverse reactions of previous treatments have not recovered to CTCAE 5.0 standard ≤ grade 1, except for grade 2 hair loss, non clinically significant and asymptomatic abnormal laboratory test values, stable hypothyroidism treated with hormone replacement therapy, and other adverse reactions that have been determined by researchers to have no safety risks.
6. Individuals who have undergone major surgical treatment, significant traumatic injury, or expected major surgery during the study treatment period within the first 4 weeks of randomization, or have long-term untreated wounds or fractures. (Note: Major surgery is defined as surgery at level 3 or above in the National Surgical Classification Catalogue 2022 edition)
7. Within the first 4 weeks of randomization, any severe (≥ CTCAE grade 3) bleeding or bleeding events occurred.
8. Uncontrolled pleural effusion and ascites with clinical significance that require repeated drainage, as well as moderate or greater amounts of pericardial effusion.
9. Individuals who have experienced arterial/venous thrombotic events within the first 6 months of randomization, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis, pulmonary embolism, or any other history of severe thromboembolism (implantable venous infusion port or catheter-related thrombosis, or superficial venous thrombosis is not considered "severe" thromboembolism).
10. Suffering from significant cardiovascular disease.
11. Brain or mental abnormalities.
12. lung disease.
13. Active or uncontrolled infections.
14. Unexplained fever>38.5 ℃ occurred during the screening period or before the first medication.
15. Patients with renal failure who require hemodialysis or peritoneal dialysis and have a history of nephrotic syndrome.
16. History of immunodeficiency, including HIV positivity or other acquired or congenital immunodeficiency diseases.
17. Patients with hypothyroidism and type 1 diabetes who are suffering from autoimmune diseases that need systemic treatment or who have received stable alternative treatment can be selected.
18. Preparing for or having previously received organ transplantation, or having a significant host transplant response, or having previously received allogeneic hematopoietic stem cell transplantation.
19. Systemic immunosuppressive therapy is required, including but not limited to: using cyclosporine, tacrolimus, etc. within the first 4 weeks of randomization, receiving high-dose glucocorticoid therapy (prednisone>30 mg/day or equivalent dose of other glucocorticoids), or receiving any other immunosuppressive therapy; Those who receive inhaled or topical corticosteroid treatment, or those who maintain a stable dose of prednisone<10 mg/day or equivalent doses of other corticosteroid systems for at least 4 weeks prior to the first administration, or those who receive steroid controlled lymphoma symptoms or prophylactic medication to prevent infusion reactions prior to the administration of the investigational drug, may be selected.
20. Known or suspected history of hemophagocytic lymphohistiocytosis (HLH).
21. Previous history of anti-tumor treatment.
22. Known to be allergic to research drug excipient components.
23. Participated in and used other anti-tumor clinical trial drugs within the first 4 weeks or 5 half lives of randomization.
24. According to the researcher's perspective, other severe, acute, or chronic medical or mental illnesses or laboratory abnormalities that may increase the risks associated with participating in the study or interfere with the interpretation of the research results.
25. It is estimated that the patient's compliance in participating in this clinical study is insufficient.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) evaluated by an independent review committee (IRC) | 2 years
  Progression free survival (PFS) evaluated by an independent review committee (IRC)

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2 years
  The percentage of complete (CR) or partial response (PR) subjects determined by IRC based on the 2014 Lugano criteria or by researchers based on the 2014 Lugano criteria and LYRIC, respectively
Complete response rate (CR rate) | 2 years
  The percentage of complete (CR) subjects determined by IRC based on the 2014 Lugano criteria or by researchers based on the 2014 Lugano criteria and LYRIC, respectively.
Progression free survival (PFS) evaluated by researchers | 2 years
  The time from randomization to researcher evaluation of disease progression or death from any cause (whichever occurs first) is determined according to the 2014 Lugano criteria and LYRIC.
Time to relief (TTR) | 2 years
  The time from randomization to first remission assessed by IRC or researchers.
Patient Outcome Report (PRO) | 2 years
  European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30), Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym) scale.
Second progression free survival (PFS2) evaluated by researchers | 2 years
  The time for the first assessment of disease progression or death from any cause (whichever occurs first) by the investigator after receiving transfer treatment or treatment allowed by the protocol, from randomization to the first IRC confirmation of disease progression, shall be determined according to the 2014 Lugano criteria and LYRIC, respectively.
The incidence and severity of adverse events (AEs) | 2 years
  The incidence and severity of adverse events (AEs), abnormal laboratory test values, and serious adverse events (SAEs).
Anti-Drug Antibodies (ADA) positivity rates | 2 years
  ADA positivity rates
Nab positivity rates | 2 years
  Nab positivity rates
Concentration of TBQ2825 in plasma | 2 years
  Concentration of TBQ2825 in plasma

CONTACTS AND LOCATIONS:
Locations (28):
- China (28):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - Sun Yet-Sen University Cancer Certer, Guangzhou, Guangdong
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Hainan General Hospital, Haikou, Hainan
  - Affiliated Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital Of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - People's Hospital of Hunan Province, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The Second Hospital Of Dalian Medical University, Dalian, Liaoning
  - Shengjing Hospital Of China Medical University, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Linyi City People Hospital, Linyi, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - People's Hospital of Tianjin, Tianjin, Tianjin Municipality
  - Tianjin Cancer Hospital Airport Hospital, Tianjin, Tianjin Municipality
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - The First People's Hospital Of Yunnan Province, Kunming, Yunnan
  - Yunan Cancer Hospital, Kunming, Yunnan